CLINICAL TRIAL: NCT03215173
Title: Fit After Baby: A Randomized Controlled Trial of a Mobile Health Intervention to Increase Postpartum Weight Loss in Women at Increased Risk for Cardiometabolic Disease
Brief Title: Fit After Baby: Increasing Postpartum Weight Loss in Women at Increased Risk for Cardiometabolic Disease
Acronym: FAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-0045
Record Dates: First submitted 2017-06-29; First posted 2017-07-12 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Cardiovascular Diseases; Diabetes; Gestational Diabetes; Preeclampsia; Gestational Hypertension; Small for Gestational Age at Delivery; Preterm Birth; Overweight and Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Diabetes, Gestational; Pre-Eclampsia; Hypertension, Pregnancy-Induced; Premature Birth; Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fit After Baby Group (Experimental): Fit After Baby mobile health lifestyle intervention to increase postpartum weight loss, increase postpartum physical activity, and improve postpartum diet.
  Interventions: Behavioral: Fit After Baby
- Text4Baby Control Group (Active Comparator): Receive text messages from the free Text4Baby program.
  Interventions: Behavioral: Text4Baby Control Group

INTERVENTIONS:
Behavioral: Fit After Baby — Mobile application
  Arms: Fit After Baby Group
Behavioral: Text4Baby Control Group — Receive free text messages
  Arms: Text4Baby Control Group

SUMMARY:
This study plans to learn more about how to increase postpartum weight loss and how to decrease risk factors for postpartum women at increased risk for diabetes and heart disease. The program is delivered using a mobile application (app) and a lifestyle coach. This mobile application is developed for women who are at higher risk for diabetes and heart disease. Women who have gestational diabetes, (diabetes during pregnancy, or GDM), gestational hypertension (high blood pressure), and/or preeclampsia (high blood pressure and protein in the urine), and/or small-for gestational-age, and/or preterm (early) delivery during their pregnancies have a higher risk for diabetes and heart disease. This mobile application was developed using the latest research studies and using the evidence-based Diabetes Prevention and Colorado Weigh programs. The goal of the program is to help women lose weight and participate in physical activity after delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45
2. Postpartum Body Mass Index (BMI): 26- 45 kg/m2 (≥24 for Asians)
3. Positive history of one or more of the following complications in most recent singleton or twin pregnancy:

   1. Gestational diabetes mellitus (by Carpenter-Coustan criteria, IADPSG (International Association of the Diabetes and Pregnancy Study Groups) criteria, or a documented clinical diagnosis). Women with a glucose value >200 mg/dL after a 50-g glucose challenge test at >12 weeks gestation will also be included.
   2. Preeclampsia (high blood pressure and proteinuria diagnosed after 20 weeks gestation)
   3. Gestational hypertension (new hypertension diagnosed after 20 weeks without proteinuria)
   4. Pre-term delivery (32-37 weeks)
   5. Small for gestational age (<10th percentile for gestational age)
4. Access to and be willing to use a wi-fi enabled iPhone (5 or higher) or iPod (5 or higher).
5. Capable of providing informed consent
6. Between 4 weeks and 16 weeks after delivery

Exclusion criteria include:

1. Personal history of Type 1 or 2 diabetes
2. Personal history of breast cancer or any other type of cancer other than a basal cell skin cancer;
3. Personal history of major chronic illness all to be assessed by the study physician for ability to participate, including:

   1. cardiovascular disease (coronary artery disease, congestive heart failure, valvular heart disease, stroke, transient ischemic attack, or intermittent claudication),
   2. kidney disease affecting kidney function severe enough to affect participation,
   3. liver disease affecting liver function severely enough to affect participation,
   4. venous or arterial thromboembolic disease,
   5. untreated adrenal insufficiency,
   6. depression requiring hospitalization within the past 6 months, or
   7. non-pregnancy related illness requiring overnight hospitalization in the past 6 months;
4. Underlying disease/treatment that might interfere with participation in/completion of the study (e.g. significant gastrointestinal conditions, major psychiatric disorders affecting the ability to participate, and others at the discretion of the study clinician);
5. Re-current pregnancy;
6. Diagnosis of diseases associated with glucose metabolism;
7. Current or planned participation in a commercial weight loss program (i.e. Jenny Craig) over the duration of the study;
8. Previous or planned bariatric surgery;
9. Taking certain prescription medications including

   1. high dose glucocorticoids,
   2. atypical antipsychotics associated with weight gain (such as risperdal (risperidone), clozapine (clozaril), olanzapine (zyprexa), quetiapine (seroquel), etc.) or
   3. weight loss medications including prescription (Qsymia, phentermine, topiramate, Belviq, Contrave, Saxenda, Orlistat), or non-prescription (Alli) medications;
10. Taking metformin or other medications known to affect glucose metabolism;
11. Other active medical problems detected by examination or laboratory testing, at the discretion of the physician;
12. Any fasting blood glucose > 126 mg/dl, any HbA1c at or above 6.5%, or any plasma glucose >200 mg/dl during the first trimester.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 82 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Change in weight loss from baseline to one year postpartum | Baseline (~6 weeks), 6 months, and 12 months
  Documentation of any change in weight at one year postpartum compared to weight at baseline, 6 weeks, 6 months and 12 months
Change in postpartum weight retention | Pre-pregnancy, 6 weeks, 6 months, and 12 months
  Documentation of any change in postpartum weight at one year postpartum compared to pre-pregnancy weight at 6 weeks, 6 months and 12 months

SECONDARY OUTCOMES:
Evaluation of Subject Satisfaction | Weekly from Baseline (~6 weeks) to 18 weeks postpartum and then at 6 months and 12 months postpartum
  Subject satisfaction will be documented using a Likert scale
Adherence to self monitoring | Daily from Baseline to 18 weeks postpartum and then at 6 months and 12 months postpartum
  Frequency
Use of app | Daily from Baseline to 12 months postpartum
  Frequency
Number of interactions with lifestyle coach | Daily from Baseline to 12 months postpartum
  Number
Change in waist circumference | Baseline to 6 months and to 12 months
  Change in cm
Change in fasting glucose | Baseline to 6 months and to 12 months
  Change in mg/dL
Change in HbA1c | Baseline to 6 months and to 12 months
  Change in %
Change in fasting insulin | Baseline to 6 months and to 12 months
  Change in fasting insulin
Change in adiponectin | Baseline to 6 months and to 12 months
  Change in adiponectin
Change in lipids | Baseline to 6 months and to 12 months
  HDL, LDL, Triglycerides
Change in blood pressure | Baseline to 6 months and to 12 months
  Change in mmHg
Change in hsCRP | Baseline to 6 months and to 12 months
  Change in hsCRP
Change in postnatal depression score | Baseline to 6 months and to 12 months
  Edinburgh Postnatal Depression Scale
Change in Physical activity | Baseline to 6 months and to 12 months
  Modified Pregnancy Physical Activity Questionnaire (PPAQ)
Change in Social Support | Baseline to 6 months and to 12 months
  Social Support for Eating Habits Survey; Social Support for Physical Activity
Change in Self-Efficacy | Baseline to 6 months and to 12 months
  Self Efficacy Survey for Diet and Exercise Behaviors
Change in Perceived Stress | Baseline to 6 months and to 12 months
  Perceived Stress Scale
Change in dietary intake | Baseline to 6 months and to 12 months
  2005 Block FFQ
Change in breastfeeding status | Baseline to 6 months and to 12 months
  Breastfeeding frequency and intensity
Change in Readiness to Change | Baseline to 6 months and to 12 months
  Readiness to Change Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jacinda Nicklas, MD, MPH, MA, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No